CLINICAL TRIAL: NCT03490344
Title: Short Course Daratumumab in Minimal Residual Disease (MRD) Positive Myeloma Patients After Induction Therapy With/Without Consolidative High Dose Chemotherapy/Autologous Stem Cell Support
Brief Title: Short Course Daratumumab in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-048
Record Dates: First submitted 2018-03-30; First posted 2018-04-06 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2023-03

CONDITIONS: Multiple Myeloma
Keywords: bony plasmacytoma; extramedullary plasmacytoma; Daratumumab; lenalidomide; Memorial Sloan Kettering Cancer Center; 18-048
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Multiple Myeloma (Experimental): Participants with MM with very good partial response (VGPR) or better after induction therapy with/without consolidative HDT/ASCT and MRD positive by bone marrow flow cytometry and MM participants who were previously MRD negative after induction and consolidation and recently (within last 3 months) turned MRD positive by bone marrow flow cytometry will be enrolled.
  Interventions: Drug: Daratumumab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Daratumumab — * Cycles 1 and 2: Daratumumab 16mg/kg weekly per cycle (28 days) as intravenous infusion (total duration: 8 weeks)
  * Cycles 3-6: Daratumumab 16mg/kg once every 2 weeks per cycle (28 days) as intravenous infusion (total duration: 16 weeks)
Drug: Lenalidomide — Lenalidomide maintenance therapy to be administered as standard treatment to all participants. This is administered as 5-15 mg daily 21-28/28 day cycle.

SUMMARY:
The purpose of this study is to test the safety of short course Daratumumab in combination with lenalidomide and to find out what effects, if any, short course Daratumumab in combination with lenalidomide has on people and their risk of multiple myeloma. The study is also designed to test the amount of remaining myeloma cells in your body after treatment with daratumumab which is known as minimal residual disease (MRD).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of Multiple Myeloma who have achieved a VGPR or better (based on best response) after induction with or without consolidation therapy/ HDT ASCT
* MRD positive at screening by flow cytometry
* Additionally, patients who were previously MRD negative after induction therapy with/without consolidative HDT/ASCT and have turned MRD positive (by flow cytometry) based on bone marrow done at screening and do not have any evidence of progressive disease are eligible
* Patients must be on standard of care lenalidomide maintenance therapy for at least 6 months at the time of study enrollment
* Patient can be receiving bisphosphonate therapy per the treating oncologist's discretion
* Creatinine clearance ≥45 ml/min using the Cockcroft-Gault method, MDRD, or CKD-EPI formula. If the calculated CrCl based on Cockcroft-Gault method, MDRD, or CKD-EPI is <45 mL/min, patient will have a 24 hr urine collection to measure CrCl.
* Age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Male or female patient who accepts and is able to use recognized effective contraception (oral contraceptives, IUCD, barrier method of contraception in conjunction with spermicidal jelly) throughout the study when relevant.
* Absolute neutrophil count (ANC) ≥1.0 x 10^9/L, hemoglobin ≥8 g/dL, and platelet count ≥75 x 10^9/L. No transfusion or growth factor support for one week prior to labs.
* Adequate hepatic function, with bilirubin < 1.5 x the ULN, and AST and ALT < 2.5 x ULN

Exclusion Criteria:

* Patients with a diagnosis of MM not achieving a VGPR or better to the most recent therapy.
* Patients with a diagnosis of MM who are MRD Negative by flow cytometry
* Patients must not have measurable disease at the time of enrollment. Measurable disease is defined as follows

  * Serum monoclonal protein > 0.5 gm/dL
  * Urine monoclonal protein > 200 mg/24 hours
  * Involved serum free light chain > 10 mg/dL
* Pregnant or lactating females
* Uncontrolled hypertension or diabetes
* Has significant cardiovascular disease with NYHA Class III or IV symptoms, or hypertrophic cardiomegaly, or restrictive cardiomegaly, or myocardial infarction within 3 months prior to enrollment, or unstable angina, or unstable arrhythmia
* Uncontrolled intercurrent illness including but not limited to active infection or psychiatric illness/social situations that would compromise compliance of study requirements
* Active infection requiring treatment within two weeks prior to first dose
* Contraindication to any concomitant medication, including antivirals, anticoagulation prophylaxis, tumor lysis prophylaxis, or hydration given prior to therapy
* Major surgery within 1 month prior to enrollment
* Previous therapy with daratumumab or other anti-CD38 monoclonal antibodies
* History of other malignancy (apart from basal cell carcinoma of the skin, or in situ cervix carcinoma) except if the patient has been free of symptoms and without active therapy during at least 5 years
* Active hepatitis B or C infection
* Subject is:

  * seropositive for human immunodeficiency virus (HIV)
  * seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR. seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sham Mailankody, MBBS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memoral Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memoral Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memoral Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://mskcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants With Multiple Myeloma
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Multiple Myeloma
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 65 [47 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With MRD Negativity by the Completion of 6 Months of Daratumumab Therapy
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Multiple Myeloma
Number analyzed (Participants) | 10
Participants
  Conversion from MRD-negativity to MRD-positivity | 6
  Persistent MRD-positivity | 4

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Participants With Multiple Myeloma
All-Cause Mortality (participants affected / at risk) | 3/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Multiple Myeloma (N=10)
Death NOS (General disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/44/NCT03490344/Prot_SAP_000.pdf